CLINICAL TRIAL: NCT01057654
Title: A Stable-isotope Study in Healthy Normolipidemic Volunteers Comparing the Mechanisms of Action of Lifibrol and Pravastatin
Brief Title: A Study Comparing the Mechanisms of Action of Lifibrol and Pravastatin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Heiner K. Berthold, MD, PhD, Dept. of Clinical Pharmacology, University of Bonn, Germany
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: LIF293/95apoB
Record Dates: First submitted 2010-01-26; First posted 2010-01-27 (Estimated); Last update posted 2010-01-27 (Estimated); Status verified 2010-01

CONDITIONS: Hypercholesterolemia; Hyperlipoproteinemia
Keywords: Cholesterol
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipoproteinemias | interventions — Pravastatin; lifibrol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lifibrol (Experimental): Lifibrol (K12.148; 4-(4'-tert. butylphenyl)-1-(4'-carboxyphenoxy)-2-butanol) given as a 600 mg film-coated tablet
  Interventions: Drug: Lifibrol
- Pravastatin (Active Comparator): Pravastatin 40 mg per day
  Interventions: Drug: Pravastatin

INTERVENTIONS:
Drug: Pravastatin — Pravastatin 40 mg
  Arms: Pravastatin
Drug: Lifibrol — Lifibrol (K12.148; 4-(4'-tert. butylphenyl)-1-(4'-carboxyphenoxy)-2-butanol) given as a 600 mg film-coated tablet
  Arms: Lifibrol

SUMMARY:
Lifibrol is a new lipid-lowering drug which lowers cholesterol to an extent in the order of magnitude of the statins. The mechanism of action of this compound is different from the one of statins but remains unknown. The current study will investigate the mechanism of action using stable-isotope turnover methods. The study will be done in healthy male volunteers.

DETAILED DESCRIPTION:
Elevated lipoprotein concentrations are a major risk factor for the development of atherosclerotic cardiovascular disease. Effective reduction of low density lipoprotein (LDL)-cholesterol concentrations has been shown to greatly reduce this risk. The most widely used lipid-lowering agents are the 3-hydroxy-3-methylglutaryl coenzyme A (HMG-CoA) reductase inhibitors (statins), which have been shown to reduce morbidity and mortality from coronary heart disease (CHD) in large prospective clinical trials. However, despite significant LDL-C reduction approximately 70% of the events are still not avoided and the search for improved or alternative lipid-modifying drug therapies continuous. HDL-C has been addressed as a potential modifiable target for decreasing this residual risk, since a low HDL-C concentration is an acknowledged independent risk factor for CHD. However, recent studies showed that an increase in HDL-C concentrations was surprisingly not associated with a decrease in atherosclerosis, but with a possible increase. Therefore it seems that not the concentrations of HDL-C should be targeted but HDL function in reverse cholesterol transport.

Lifibrol is a lipid-modifying drug which has been shown to improve HDL particle flux via increased apoA-I production, while not having HDL-raising properties. Furthermore, it decreases dose-dependently LDL-C by up to 40%. It is of major interest to clarify the, apparently unique, mechanisms of action of a compound, whose LDL-lowering effects are comparable in magnitude to the ones of statins.

The mechanisms of lifibrol's LDL-lowering effects are not completely clarified. There is evidence suggesting that it increases hepatic LDL receptor expression by a sterol-independent mechanism, i.e. not through a reduction in cholesterol synthesis, the mechanism of action of statins. ApoB turnover studies have indicated that increased catabolism of LDL rather than a decrease in hepatic apoB production may be responsible for its cholesterol-lowering effects. Since apoB metabolism and cholesterol synthesis are closely related, we designed a study to investigate the effects of lifibrol on the metabolism of apoB-100-containing lipoproteins and on endogenous sterol synthesis in parallel, using stable isotope methods. In addition, since lifibrol may inhibit cholesterol synthesis at steps earlier than HMG-CoA reductase, we investigated [13C]acetate catabolism analyzing 13CO2 appearance in breath. The HMG-CoA-reductase inhibitor pravastatin was used as comparator, since its mode of action is well characterized. The principle questions addressed were (i) whether lifibrol exerts its cholesterol-lowering effects through decreased synthesis/enhanced catabolism of apoB-100-containing lipoproteins or through inhibition of sterol de novo synthesis and (ii) whether these effects are interrelated.

ELIGIBILITY:
Inclusion Criteria:

* male volunteers
* 18 to 35 years old
* good clinical condition
* normal eating habits
* mental abilities to be able to understand the study procedures
* written informed consent

Exclusion Criteria:

* relevant pathological findings in the baseline examination
* known allergic predisposition
* concomitant drugs
* alcohol or nicotine abuse
* participation in other clinical trials in the last 30 days

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 1996-01; Primary Completion 1996-04 (Actual); Study Completion 1998-06 (Actual)

PRIMARY OUTCOMES:
LDL cholesterol lowering | 4 weeks

SECONDARY OUTCOMES:
Changes in other lipoprotein concentrations | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Heiner K. Berthold, Professor, Principal Investigator — University of Bonn
Locations (1):
- Dept. of Clinical Pharmacology, University of Bonn, Bonn, Germany